CLINICAL TRIAL: NCT00071110
Title: Electroacupuncture for Major Depression: A Pilot Study
Brief Title: Electroacupuncture for Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT001218-01A1 (NIH)
Record Dates: First submitted 2003-10-10; First posted 2003-10-15 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2009-12

CONDITIONS: Depression; Depressive Disorder
Keywords: Acupuncture; Electroacupuncture; Alternative therapy
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Electroacupuncture; salicylhydroxamic acid

ARMS (2):
- 1 (Experimental): Electroacupuncture (EA).
  Interventions: Procedure: Electroacupuncture
- 2 (Placebo Comparator): Sham
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Electroacupuncture — For subjects randomized to EA, needles were placed at points GV-20-on the crown of the head and yin tang-on the midline of the forehead roughly at the glabella and treated with electrical stimulation. 30 mm x 0.22 mm sterile stainless steel needles were placed obliquely to a depth of approximately 10 mm and were connected to face-microelectrodes which were connected to the Pantheon Research PENS-Electrostimulator. Electricity was provided at a frequency of 2 Hz and set to a voltage which resulted in the perception of a mild intensity stimulation.
  Arms: 1
Procedure: Sham — For subjects randomized to SA, two needles were placed laterally on the scalp, 3 cuns superior to the temporal attachment of the helix of the ear. This point was selected as it does not correspond to any specific meridian acupuncture point. A disabled electrical cable was connected to the needles and the electrostimulator, with light blinking at 2 Hz but no electrical stimulation provided.
  Arms: 2

SUMMARY:
This study will compare the safety, efficacy, and tolerability of electroacupuncture (EA) and sham electroacupuncture (SA) for the treatment of major depression.

DETAILED DESCRIPTION:
Major depression is a common and serious mental illness. It is associated with a markedly lower quality of life, significant functional impairment, and premature death due to suicide or comorbid physical illness. Over the past 50 years, effective and safe treatments for major depression have been developed, including antidepressant pharmacotherapy, psychotherapy, and electroconvulsive therapy. However, many Americans who suffer from a depressive disorder either do not elect to receive one of these conventional treatments or do not complete an adequate course of treatment. A growing number of Americans with depression are choosing to be treated with complementary and alternative therapies. Acupuncture, in particular, is increasingly being used to treat depression even though only limited data support its safety and efficacy.

This study will use a randomized parallel-group design to compare the safety, efficacy, and tolerability of electroacupuncture (EA) and sham electroacupuncture (SA) for the treatment of major depression. Over a 15-month period, 60 adult outpatients with a major depressive disorder of mild or moderate severity (as defined by the DSM-IV) will be randomized to either 12 sessions of EA or SA to be provided over 6 weeks. Safety and symptomatic improvement (as measured with the Hamilton Rating Scale for Depression [HRSD]) will constitute the primary outcome measures. Tolerability and functional improvement will constitute secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Meet SCID criteria for a Major Depressive Disorder (Single or Recurrent) with a current major depressive episode of mild or moderate severity
* Significant symptoms of depression (HRSD > 14)
* Ability to communicate in English
* Give informed consent in accordance with local IRB regulations

Exclusion Criteria:

* Personal physician's recommendation against enrollment because the patient is physically unstable or for other reasons
* Having been treated with acupuncture for any condition
* History of seizure disorder or significant risk factors for a seizure disorder (e.g., history of brain trauma, recent stroke, or brain tumor)
* Need to remain on antidepressant or other psychotropic medications
* Absence of depressive symptoms severe enough (i.e., HRSD < 14) at the baseline assessments
* Significant cognitive impairment, as assessed by a total score on the MMSE < 25. A recommendation for referral to a neurologist or a psychiatrist will be made to the patient in these cases.
* Chronic major depression (i.e, duration of 2 years or longer) A recommendation for referral to a psychiatrist will be made in these cases.
* Major depressive episode severe or severe with psychotic features (as per DSM-IV/SCID) or with acutely suicidality. A recommendation for psychiatric referral will be made in these cases. Bipolar disorder, psychotic features, or a psychotic disorder (specifically: schizophrenia, delusional disorder, or schizoaffective disorder). A recommendation for psychiatric referral will be made in these cases.
* Met criteria for a diagnosis of alcohol substance abuse or dependence within the past six months. A recommendation for referral to a mental health professional will be made in these cases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit H Mulsant, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside, Center for Complementary Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Andreescu C, Glick RM, Emeremni CA, Houck PR, Mulsant BH. Acupuncture for the treatment of major depressive disorder: a randomized controlled trial. J Clin Psychiatry. 2011 Aug;72(8):1129-35. doi: 10.4088/JCP.10m06105. Epub 2011 May 3. PMID 21672495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 Participants were recruited from March 2004 - May 2007 at the UPMC Shadyside Center for Complementary Medicine.
Pre-assignment Details: Twenty-nine subjects were randomized to Sham and 28 to Electroacupuncture.
Groups:
- Electroacupuncture (EA): Needles placed at traditional meridian locations, GV-20 (on the crown of the head) and yin tang (in the midline of the forehead roughly at the glabella) and treated with electrical stimulation.
- Sham Acupuncture (SA): Needles placed laterally on the scalp, not corresponding to any traditional meridians. No electrical stimulation delivered.
Period: Overall Study
Arm/Group | Electroacupuncture (EA) | Sham Acupuncture (SA)
Started | 28 | 29
Completed | 28 | 25
Not Completed | 0 | 4
Not completed — Protocol Violation | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electroacupuncture (EA) | Sham Acupuncture (SA) | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 28 | 25 | 53.0
  >=65 years | 0 | 4 | 4.0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.04 (11.32) | 48.86 (13.12) | 47.47 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39.0
  Male | 7 | 11 | 18.0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57.0

OUTCOME MEASURES:

1. Primary Outcome: Antidepressant Response, Defined as a Hamilton Depression Rating Scale Score Relative Decrease of 50 % or More and a Final Score < 10
Description: Number of participants whose Hamilton Depression Rating Scale score decreased at least 50% and had a final score less than 10. Minimum score = 0 (best). Maximum score = 52 (worst). The 17 item scale assesses depression symptoms, including Depressed Mood, Feelings of Guilt, Suicidal Ideation, Insomnia, Anxiety, Weight Change, and Insight.
Time Frame: Change from Baseline to Post-Intervention Endpoint
Population: ITT, excluding the first four sham acupuncture subjects, whom the primary acupuncturist erred in treating. Although he correctly used the sham electricity procedure, for these subjects he placed needles in the verum electroacupuncture points of GV-20 and Yin tang.
Measure: Number; unit: participants
Arm/Group | Electroacupuncture (EA) | Sham Acupuncture (SA)
Number analyzed (Participants) | 28 | 25
participants | 11 | 11

2. Secondary Outcome: Change in Functioning and Health-related Quality of Life as Rated by the Medical Outcomes Survey-Version 1 (MOS-36) Physical Component Score (MOSPCS)
Description: Mean change in scores on the Medical Outcomes Survey-Version 1 (MOS-36) PHYSICAL Component Score (MOSPCS) from baseline to post-intervention across treatment group. Minimum Score = 0 (worse); Maximum Score = 100 (better), Normed to be at 50 on a control population. Positive Mean Change scores indicate improvement (an increase in scale score/better).
Time Frame: Mean Change from Baseline to Post-Intervention Endpoint
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Electroacupuncture (EA) | Sham Acupuncture (SA)
Number analyzed (Participants) | 28 | 25
Units on a scale | 0.54 (6.92) | -1.65 (7.98)
Statistical Analysis 1: Comparison: Electroacupuncture (EA) vs Sham Acupuncture (SA); Test type: Superiority or Other; p = 0.32, t-test, 2 sided — Statistic (t): -1.00

3. Secondary Outcome: Change in Functioning and Health-related Quality of Life as Rated by the Medical Outcomes Survey-Version 1 (MOS-36) Mental Component Score (MOSMCS)
Description: Mean change in scores on the Medical Outcomes Survey-Version 1 (MOS-36) Mental Component Score (MOSMCS) from baseline to post-intervention across treatment group. Minimum Score = 0 (worse); Maximum Score = 100 (better) , Normed to be at 50 on a control population. Positive Mean Change scores indicate improvement (an increase in scale score).
Time Frame: Mean Change from Baseline to Post-Intervention Endpoint
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Electroacupuncture (EA) | Sham Acupuncture (SA)
Number analyzed (Participants) | 28 | 25
Units on a scale | 6.23 (13.62) | 14.12 (17.54)
Statistical Analysis 1: Comparison: Electroacupuncture (EA) vs Sham Acupuncture (SA); Test type: Superiority or Other; p = 0.09, t-test, 2 sided — Statistic (t): 1.56

4. Secondary Outcome: Change in Functioning and Health-related Quality of Life as Rated by the Medical Outcomes Survey-Version 1 (MOS-36) Bodily Pain Index (MOSBPI)
Description: Mean change in scores on the Medical Outcomes Survey-Version 1 (MOS-36) Bodily Pain Index (MOSBPI) from baseline to post-intervention across treatment group. Minimum Score = 0 (more); Maximum Score = 100 (less). Positive Mean Change scores indicate improvement (an increase in scale score/less pain).
Time Frame: Mean Change from Baseline to Post-Intervention Endpoint
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Electroacupuncture (EA) | Sham Acupuncture (SA)
Number analyzed (Participants) | 28 | 25
Units on a scale | -1.04 (18.27) | 6.81 (19.70)
Statistical Analysis 1: Comparison: Electroacupuncture (EA) vs Sham Acupuncture (SA); Test type: Superiority or Other; p = 0.17, t-test, 2 sided — Statistic (t): 1.40

ADVERSE EVENTS:
Time Frame: Weekly assessments from Baseline to Post-Intervention endpoint
Description: SEMI-STRUCTURED INTERVIEW FOR THE Udvalg Fur Kliniske Undersogesler (UKU) SIDE EFFECTS RATING SCALE From the University of Pittsburgh. Adapted by Tracy Flynn, M.S. Ed. and Benoit H. Mulsant, M.D. from: Lingjaerde O, Ahlfors UG, Bech P, Dencker SJ, Elgen K (1987). The UKU side effect rating scale. Acta Psychitr Scand 334(Suppl): 1-100
Arm/Group | Electroacupuncture (EA) | Sham Acupuncture (SA)
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 23/28 | 25/29
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Electroacupuncture (EA) (N=28) | Sham Acupuncture (SA) (N=29)
CONCENTRATION DIFFICULTIES (Psychiatric disorders) | 0 | 3 — Udvalg Fur Kliniske Undersogesler (UKU) Question 1: CONCENTRATION DIFFICULTIES: difficulties in ability to concentrate, to collect one's thoughts, or to sustain one's attention.
ASTHENIA / LASSITUDE / INCREASED FATIGUABILITY (Psychiatric disorders) | 1 | 2 — Udvalg Fur Kliniske Undersogesler (UKU) Question 2: ASTHENIA / LASSITUDE / INCREASED FATIGUABILITY: the patient's experience of lassitude and lack of endurance. The assessment is based upon the patient's reported statements.
SLEEPINESS / SEDATION (Psychiatric disorders) | 1 | 1 — Udvalg Fur Kliniske Undersogesler (UKU) Question 3: SLEEPINESS / SEDATION: diminished ability to stay awake during the day. The assessment is based on clinical signs during the interview.
FAILING MEMORY (Psychiatric disorders) | 1 | 1 — Udvalg Fur Kliniske Undersogesler (UKU) Q4-FAILING MEMORY: impaired memory. Assessment should be independent of any concentration difficulties.
TENSION / INNER UNREST (Psychiatric disorders) | 1 | 3 — Udvalg Fur Kliniske Undersogesler (UKU) Q6-TENSION / INNER UNREST: inability to relax, nervous restlessness. This item is to be assessed on the basis of the patient's experience and must be distinguished from motor akathesia (Q16).
INCREASED DURATION OF SLEEP: (Psychiatric disorders) | 3 | 4 — Udvalg Fur Kliniske Undersogesler (UKU) Q7-INCREASED DURATION OF SLEEP: this should be assessed on the basis of the average of sleep over the three preceding nights. The assessment is to be made in relation to the patient's usual pre-illness state.
REDUCED DURATION OF SLEEP: (Psychiatric disorders) | 7 | 7 — Udvalg Fur Kliniske Undersogesler (UKU) Q8-REDUCED DURATION OF SLEEP: should be assessed on the basis of the average of sleep over the three preceding nights. The assessment is to be made in relation to the patient's usual pre-illness state.
INCREASED DREAM ACTIVITY (Psychiatric disorders) | 9 | 12 — Udvalg Fur Kliniske Undersogesler (UKU) Q9-INCREASED DREAM ACTIVITY: should be assessed independently of dream content and based on the average of sleep over the preceding nights in relation to the usual pre-illness dream activity.
EMOTIONAL INDIFFERENCE (Psychiatric disorders) | 2 | 2 — Udvalg Fur Kliniske Undersogesler (UKU) Q10-EMOTIONAL INDIFFERENCE: a diminution of the patient's empathy, leading to apathy.
TREMOR (Nervous system disorders) | 0 | 1 — UKU Q15-TREMOR: this item comprises all forms of tremor.
PARATHESIAS (Nervous system disorders) | 0 | 1 — UKU Q18-PARATHESIAS: pricking, creeping, or burning sensations in the skin.
HEADACHE (Nervous system disorders) | 8 | 4 — UKU Q19-HEADACHE: on the scoring sheet headache is classified as (a) tension headache, (b) migraine, or (c) other forms of headache
ACCOMMODATION DISTURBANCES (Nervous system disorders) | 0 | 1 — UKU Q20-ACCOMMODATION DISTURBANCES: difficulty in seeing clearly or distinctly at close quarters (with or without glasses), whereas the patient sees clearly at a long distance (w/glasses if necessary)
NAUSEA / VOMITING (Gastrointestinal disorders) | 7 | 3 — UKU Q23-NAUSEA / VOMITING: to be recorded on the basis of the last 3 days.
DIARRHEA (Gastrointestinal disorders) | 1 | 1 — UKU Q24-DIARRHEA: increased frequency and or thinner consistency of feces.
CONSTIPATION (Gastrointestinal disorders) | 0 | 3 — UKU Q25-CONSTIPATION: reduced frequency of defection and/or thicker consistency of feces.
MICTURITION DISTURBANCES (Renal and urinary disorders) | 0 | 1 — UKU Q26-MICTURITION DISTURBANCES: feeling of difficulty in starting and or resistance to micturition, weaker stream and/or increased time of micturition. Should be assessed on the basis of the last 3 days.
ORTHOSTATIC DIZZINESS (Nervous system disorders) | 3 | 3 — UKU Q28-ORTHOSTATIC DIZZINESS: feeling of weakness, everything going black, buzzing in the ears, increasing tendency to faint when changing from supine or sitting position to upright position.
PALPITATIONS / TACHYCARDIA (Cardiac disorders) | 2 | 1 — UKU Q29-PALPITATIONS / TACHYCARDIA: palpitation, feeling of rapid, strong and /or irregular heartbeats.
INCREASED TENDENCY TO SWEATING (Skin and subcutaneous tissue disorders) | 3 | 1 — UKU Q30-INCREASED TENDENCY TO SWEATING: localized to the whole body, not only palms and soles of the foot.
RASH (Skin and subcutaneous tissue disorders) | 1 | 2 — UKU Q31-RASH: for scoring, the types of rashes are classified as (a) morbilliform, (b) petechial, (c) urticarial, (d) psoriataic, and (e) cannot be classified.
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 1
PHOTOSENSITIVITY (Skin and subcutaneous tissue disorders) | 2 | 2 — UKU Q33-PHOTOSENSITIVITY: increased sensitivity to sunlight.
WEIGHT LOSS (Metabolism and nutrition disorders) | 0 | 2
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 1 — UKU Q37-(Menstruating females only) MENORRHAGIA: hypermenorrhea, polymenorrhea, or metrorrhagia during the last 3 months (or since last assessment).
DIMINISHED SEXUAL DESIRE (Reproductive system and breast disorders) | 3 | 5
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 1 — UKU Q43-(Sexually active males only) ERECTILE DYSFUNCTION: difficulty in attainting or maintaining an erection.
EJACULATORY DYSFUNCTION (Reproductive system and breast disorders) | 0 | 1 — UKU Q44-(Sexually active males only) EJACULATORY DYSFUNCTION: dysfunction of the patient's ability to control ejaculation. Includes (a) premature or (b) delayed ejaculation.
ORGASMIC DYSFUNCTION (Reproductive system and breast disorders) | 7 | 4 — UKU Q45-(Sexually active females and males) ORGASMIC DYSFUNCTION: difficulty in obtaining and experiencing satisfactory orgasm.
DRY VAGINA (Reproductive system and breast disorders) | 1 | 0 — Q46-(Sexually active females only) DRY VAGINA: dryness of vagina with sexual stimulation.

LIMITATIONS AND CAVEATS:
Four participants were excluded from the analyses because of a protocol violation. In the Sham Acupuncture group, the acupuncturist placed unelectrified needles in GV-20 and Yin tang points instead of placing them laterally.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No